CLINICAL TRIAL: NCT05308979
Title: Intradetrusor Botulinum Toxin A for OAB Via 1 Versus 10 Injections: A Randomized Clinical Trial
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, Irvine (Other)
Collaborators: Kaiser Permanente (Other); St. Joseph Hospital of Orange (Other)
Responsible Party: Principal Investigator, Carly Ann Crowder, Fellow Physician, PI, University of California, Irvine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 309
Record Dates: First submitted 2022-03-15; First posted 2022-04-04 (Actual); Results first posted 2025-02-14 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Overactive Bladder; Urinary Urge Incontinence; Overactive Bladder Syndrome; Urinary Incontinence, Urge; Urge Incontinence; Urinary Urgency; Urinary Frequency
MeSH Terms: conditions — Urinary Bladder, Overactive; Urinary Incontinence, Urge | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Intervention Model Description: Parallel study with 2 arms, 1:1 randomization
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- 1 Injection Site (Experimental): 100u Botox® injected at one intradetrusor site
  Interventions: Drug: OnabotulinumtoxinA 100 UNT [Botox]
- 10 Injection Sites (Active Comparator): 100u Botox® injected at 10 intradetrusor sites
  Interventions: Drug: OnabotulinumtoxinA 100 UNT [Botox]

INTERVENTIONS:
Drug: OnabotulinumtoxinA 100 UNT [Botox] — Intradetrusor (Bladder) Botox Injection at 1 vs 10 injection sites

SUMMARY:
Patients with either overactive bladder (OAB) or urgency urinary incontinence (UUI) with be randomized (like a flip of a coin) to receive 100 units of bladder Botox® at either one injection site or ten injection sites. Efficacy and patient satisfaction will be measured by questionnaires.

DETAILED DESCRIPTION:
Intradetrusor (bladder) Botulinum toxin A (BTA or Botox®) is a well-established treatment for urinary urgency incontinence (UUI).[1,2] While this treatment's efficacy in comparison to alternative therapies including anticholinergic medications and sacral neuromodulation for treatment of UUI has been studied, the ideal number of injection sites within the bladder has not been well established. [3,4] Intradetrusor BTA injections are often completed as an office procedure while the patient is awake. Each injection site can cause discomfort for the patient during the procedure. Urinary tract infection and urinary retention are risks associated with this procedure and could potentially be related to number of injection sites. Currently, there is a lack of information in the literature regarding the optimal number of intravesical BTA injection sites.

Prior studies evaluated efficacy using 100u BTA spread across 20 injections sites, however current practices at local institutions safely use 10 injections sites based on studies showing similar effect and adverse event profiles between use of 10, 20, and 40 injection sites.[5,6] Research using animal models has shown diffuse distribution of BTA within the entire detrusor muscle after just a single BTA injection at one site.[7] This has been corroborated in human studies.[8] A recently published observational pilot study shows promise for single site intradetrusor Botox® injection as it reported a lower rate of urinary retention and similar durability.[9] Similar clinical efficacy with only one to three intravesical BTA injection[s] has also been reported.[10]

In this study, participants will be randomized to receive 100u BTA via intradetrusor injection at one injection site (experimental) versus 10 injection sites (control). Investigators hypothesize that one injection will have similar efficacy to multiple injections and potentially better tolerability and patient satisfaction, due to decreased procedure time and less pain, along with potential for lower adverse event rates, specifically urinary retention and urinary tract infections.

ELIGIBILITY:
Inclusion Criteria:

* Female
* 18 years old or greater
* Diagnosis of overactive bladder (urinary urgency or frequency, OAB) or urinary urgency incontinence (UUI)

Exclusion Criteria:

* Have a diagnosis of neurogenic bladder
* Received intravesical botox injections within prior 6 months
* Current treatment with either: SNM, PTNS, or OAB medications - need wash out as below
* SNM - turn device off for at least 2 weeks prior to procedure, off during 3-month follow up window
* PTNS - no treatments within 2 weeks of start, none during 3-month post-procedure follow up window
* OAB meds - 2 week wash out period prior to injection, none during 3-month post-procedure follow up window
* Currently pregnant or trying to get pregnant
* Contraindications to Botox® - hypersensitivity to Botox®, inability to self-catheterize/refusal to have indwelling catheter
* Have a UTI (can enroll after treatment)
* Have urinary retention (PVR>150cc on two occasions)
* Do not speak English or Spanish

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carly Crowder, MD, Principal Investigator — UC Irvine; Taylor Brueseke, MD, Study Director — UC Irvine; Felicia Lane, MD, Study Chair — UC Irvine
Locations (1):
- University of California Irvine Medical Center, Orange, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brubaker L, Richter HE, Visco A, Mahajan S, Nygaard I, Braun TM, Barber MD, Menefee S, Schaffer J, Weber AM, Wei J; Pelvic Floor Disorders Network. Refractory idiopathic urge urinary incontinence and botulinum A injection. J Urol. 2008 Jul;180(1):217-22. doi: 10.1016/j.juro.2008.03.028. Epub 2008 May 21. PMID 18499184
- [Background] Chapple C, Sievert KD, MacDiarmid S, Khullar V, Radziszewski P, Nardo C, Thompson C, Zhou J, Haag-Molkenteller C. OnabotulinumtoxinA 100 U significantly improves all idiopathic overactive bladder symptoms and quality of life in patients with overactive bladder and urinary incontinence: a randomised, double-blind, placebo-controlled trial. Eur Urol. 2013 Aug;64(2):249-56. doi: 10.1016/j.eururo.2013.04.001. Epub 2013 Apr 10. PMID 23608668
- [Background] Visco AG, Brubaker L, Richter HE, Nygaard I, Paraiso MF, Menefee SA, Schaffer J, Lowder J, Khandwala S, Sirls L, Spino C, Nolen TL, Wallace D, Meikle SF; Pelvic Floor Disorders Network. Anticholinergic therapy vs. onabotulinumtoxina for urgency urinary incontinence. N Engl J Med. 2012 Nov 8;367(19):1803-13. doi: 10.1056/NEJMoa1208872. Epub 2012 Oct 4. PMID 23036134
- [Background] Amundsen CL, Richter HE, Menefee SA, Komesu YM, Arya LA, Gregory WT, Myers DL, Zyczynski HM, Vasavada S, Nolen TL, Wallace D, Meikle SF. OnabotulinumtoxinA vs Sacral Neuromodulation on Refractory Urgency Urinary Incontinence in Women: A Randomized Clinical Trial. JAMA. 2016 Oct 4;316(13):1366-1374. doi: 10.1001/jama.2016.14617. PMID 27701661
- [Background] Nitti VW, Dmochowski R, Herschorn S, Sand P, Thompson C, Nardo C, Yan X, Haag-Molkenteller C; EMBARK Study Group. OnabotulinumtoxinA for the treatment of patients with overactive bladder and urinary incontinence: results of a phase 3, randomized, placebo controlled trial. J Urol. 2013 Jun;189(6):2186-93. doi: 10.1016/j.juro.2012.12.022. Epub 2012 Dec 14. PMID 23246476
- [Background] Liao CH, Chen SF, Kuo HC. Different number of intravesical onabotulinumtoxinA injections for patients with refractory detrusor overactivity do not affect treatment outcome: A prospective randomized comparative study. Neurourol Urodyn. 2016 Aug;35(6):717-23. doi: 10.1002/nau.22780. Epub 2015 Apr 24. PMID 25914349
- [Background] Coelho A, Cruz F, Cruz CD, Avelino A. Spread of onabotulinumtoxinA after bladder injection. Experimental study using the distribution of cleaved SNAP-25 as the marker of the toxin action. Eur Urol. 2012 Jun;61(6):1178-84. doi: 10.1016/j.eururo.2012.01.046. Epub 2012 Feb 1. PMID 22306320
- [Background] Mehnert U, Boy S, Schmid M, Reitz A, von Hessling A, Hodler J, Schurch B. A morphological evaluation of botulinum neurotoxin A injections into the detrusor muscle using magnetic resonance imaging. World J Urol. 2009 Jun;27(3):397-403. doi: 10.1007/s00345-008-0362-0. Epub 2009 Jan 15. PMID 19145439
- [Background] Ton J, Downing P, Versi E, van Uem S, Ephraim S, Murphy M, Lucente V. Outcomes of a single trigone-only vs. 20 trigone-sparing injections of OnabotulinumtoxinA for refractory overactive bladder (OAB). Int Urol Nephrol. 2021 Jun;53(6):1067-1072. doi: 10.1007/s11255-021-02802-0. Epub 2021 Mar 19. PMID 33742316
- [Background] Avallone MA, Sack BS, El-Arabi A, Guralnick ML, O'Connor RC. Less is more-A pilot study evaluating one to three intradetrusor sites for injection of OnabotulinumtoxinA for neurogenic and idiopathic detrusor overactivity. Neurourol Urodyn. 2017 Apr;36(4):1104-1107. doi: 10.1002/nau.23052. Epub 2016 Jun 10. PMID 27283922

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 1 Injection Site | 10 Injection Sites
Started | 58 | 58
Completed | 44 | 45
Not Completed | 14 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1 Injection Site | 10 Injection Sites | Total
Number analyzed (Participants) | 58 | 58 | 116
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.9 (10.72) | 68 (11.34) | 68 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58 | 58 | 116
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 4 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 38 | 35 | 73
  More than one race | 14 | 18 | 32
  Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change in Overactive Bladder Questionnaire Long Form Score (Symptoms Severity Sub-scale)(OAB-Q LF)
Description: Participants will be asked to Overactive Bladder Questionnaire Long Form prior to receiving the Botox procedure. The OAB-Q LF symptom severity sub-scale score will be compared prior to procedure and again to score at 3 weeks after procedure.
  The OAB-q Symptom Severity Score will be computed at baseline and 3 weeks (and 3 months) using the standard scoring algorithm. Minimum value of symptom severity subscale is 8, maximum is 48. A higher score means worse symptoms. A lower score means less symptoms.
Time Frame: change from baseline OAB-Q score to 3 wk post-procedure score
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1 Injection Site | 10 Injection Sites
Number analyzed (Participants) | 58 | 58
units on a scale | -31.2 (26.25) | -39.5 (24.92)

2. Secondary Outcome: Change in Overactive Bladder Questionnaire Long Form Score (Symptoms Severity Sub-scale)(OAB-Q LF)
Description: Participants will be asked to complete Overactive Bladder Questionnaire Long Form prior to receiving the Botox procedure. The OAB-Q LF symptom severity sub-scale score will be compared prior to procedure and again to score at 3 months after procedure.
  The OAB-q Symptom Severity Score will be computed at baseline and 3 weeks (and 3 months) using the standard scoring algorithm. Minimum value of symptom severity subscale is 8, maximum is 48. A higher score means worse symptoms. A lower score means less symptoms.
Time Frame: comparison of baseline OAB-Q score to 3 month post-procedure score
Reporting Status: Not Posted

3. Secondary Outcome: Post-void Residual (PVR)
Description: A PVR will be collected via either urethral catheterization or bladder scan (ultrasound in clinic) at 3 weeks post-procedure as a marker of urinary retention. The PVRs will be compared between study and control groups
Time Frame: PVR collected at 3 wk post-procedure
Reporting Status: Not Posted

4. Secondary Outcome: Number of Participants With Urinary Tract Infection (UTI)
Description: Urine culture will be sent for any patient with urinary tract infections symptoms (eg: worsening urgency, frequency, dysuria).
Time Frame: anytime after procedure, until at least 3 months post-procedure.
Reporting Status: Not Posted

5. Secondary Outcome: Patient Global Impression - Improvement (PGI-I)
Description: Participants will complete PGI-I Questionnaire at 3 months after procedure. The minimum value is 1 (very much better) and maximum value score is 7 (very much worse). A higher score indicates worse symptoms. A lower score indicates better symptoms or more improvement.
Time Frame: 3 months after botox procedure
Reporting Status: Not Posted

6. Secondary Outcome: Visual Analogue Scale (VAS) - Pain
Description: Participants will complete VAS-pain immediately post-procedure as a pain and tolerability assessment
Time Frame: immediately after procedure
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | 1 Injection Site | 10 Injection Sites
All-Cause Mortality (participants affected / at risk) | 0/58 | 0/58
Serious Adverse Events (participants affected / at risk) | 0/58 | 0/58
Other Adverse Events (participants affected / at risk) | 0/58 | 0/58

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-09): https://cdn.clinicaltrials.gov/large-docs/79/NCT05308979/Prot_SAP_000.pdf